CLINICAL TRIAL: NCT03203824
Title: The Effects of Dark Chocolate (70% Cacao) on EEG Brain Waves in Vigorously Active Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Georgia Hodgkin, EdD, Professor, Loma Linda University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 5170184
Record Dates: First submitted 2017-06-26; First posted 2017-06-29 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dark chocolate (Experimental): Three EEG measurements will be recorded: 1) at baseline, 2) during visualization of rest for one minute, and 3) during visualization of usual vigorous exercise for one minute. Measurements 2 and 3 will be recorded savoring dark chocolate and after fully ingesting the dark chocolate respectively.
  Interventions: Dietary Supplement: dark chocolate
- non dark chocolate (Active Comparator): three EEG measurements will be recorded: 1) at baseline, 2) during visualization of rest for one minute, and 3) during visualization of usual vigorous exercise for one minute.
  Interventions: Other: non dark chocolate

INTERVENTIONS:
Dietary Supplement: dark chocolate — Participants will be provided Parliament dark chocolate (70% cocoa) from Redlands, CA. The Parliament chocolate is made with cacao and cane sugar. Each participant will be given half a piece (1.4 g) of dark chocolate to consume for this experiment over three minutes.
  Arms: dark chocolate
Other: non dark chocolate — No dark chocolate will be given to this group during the procedures.
  Arms: non dark chocolate

SUMMARY:
The purpose of this graduate student study is to determine if ingestion of dark chocolate (70% cacao) will change brain frequencies between visualization at a state of rest and a state of exercise performance via electroencephalography (EEG) in vigorously active individuals.

DETAILED DESCRIPTION:
The procedures include: On day one, participants will fill out a dark chocolate Likert scale, physical activity assessment, and demographic questionnaire. Day two and three, on consecutive days will include, three EEG measurements will be recorded: 1) at baseline, 2) during visualization of rest for one minute, and 3) during visualization of usual vigorous exercise for one minute. The second day all three measurements will be recorded without dark chocolate (70% cacao). The third day all three measurements will be recorded again. Measurements 2 and 3 will be recorded savoring dark chocolate and after fully ingesting the dark chocolate respectively.

ELIGIBILITY:
Inclusion Criteria:

* 21-45 years of age
* vigorously active individuals, based on the General Physical Activities defined by Level of Intensity guidelines, greater than 75 minutes per week
* enjoy dark chocolate

Exclusion Criteria:

* Caffeine, sedatives, or tranquilizers within 12 hours of study
* Creatine or other performance enhancing steroid supplementation within 24 hours of study
* Ginseng supplementation within 24 hours of study
* Barbiturates within at least 36 hours of study
* Currently taking antiepileptic medications
* Any allergies, colds or sinus infections day of the study

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
EEG Wave Band Activity without dark chocolate ingestion | change from baseline to during visualization of rest for one minute
  The EEG, electroencephalogram, is a test that detects abnormalities in the brain waves or the electrical activity of the brain. During the procedure, electrodes consisting of small metal discs with thin wires are pasted onto the scalp. The electrodes detect tiny electrical charges that result from the activity in the brain cells. EEG wave band activity will be recorded from 9 cerebral cortical scalp locations: F3, Fz, F4, C3, Cz, C4, P3, Pz, and P4 using the EEG B-Alert 10X System, Carlsbad CA. Each of the brain frequencies will be measured in 5 second increments. Data collection will last no longer than 2 hours for each session.
EEG Wave Band Activity without dark chocolate ingestion | change from visualization of rest for one minute and during visualization of usual vigorous exercise for one minute.
  The EEG, electroencephalogram, is a test that detects abnormalities in the brain waves or the electrical activity of the brain. During the procedure, electrodes consisting of small metal discs with thin wires are pasted onto the scalp. The electrodes detect tiny electrical charges that result from the activity in the brain cells. EEG wave band activity will be recorded from 9 cerebral cortical scalp locations: F3, Fz, F4, C3, Cz, C4, P3, Pz, and P4 using the EEG B-Alert 10X System, Carlsbad CA. Each of the brain frequencies will be measured in 5 second increments. Data collection will last no longer than 2 hours for each session.

SECONDARY OUTCOMES:
EEG wave band activity with dark chocolate ingestion | change from baseline to during visualization of rest for one minute
  The EEG, electroencephalogram, is a test that detects abnormalities in the brain waves or the electrical activity of the brain. During the procedure, electrodes consisting of small metal discs with thin wires are pasted onto the scalp. The electrodes detect tiny electrical charges that result from the activity in the brain cells. EEG wave band activity will be recorded from 9 cerebral cortical scalp locations: F3, Fz, F4, C3, Cz, C4, P3, Pz, and P4 using the EEG B-Alert 10X System, Carlsbad CA. Each of the brain frequencies will be measured in 5 second increments. Data collection will last no longer than 2 hours for each session.
EEG wave band activity with dark chocolate ingestion | change from visualization of rest for one minute and during visualization of usual vigorous exercise for one minute.
  The EEG, electroencephalogram, is a test that detects abnormalities in the brain waves or the electrical activity of the brain. During the procedure, electrodes consisting of small metal discs with thin wires are pasted onto the scalp. The electrodes detect tiny electrical charges that result from the activity in the brain cells. EEG wave band activity will be recorded from 9 cerebral cortical scalp locations: F3, Fz, F4, C3, Cz, C4, P3, Pz, and P4 using the EEG B-Alert 10X System, Carlsbad CA. Each of the brain frequencies will be measured in 5 second increments. Data collection will last no longer than 2 hours for each session.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Hodgkin, EdD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda U, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No